CLINICAL TRIAL: NCT00435058
Title: Visual Function Changes After Intraocular Pressure Reduction Using Antiglaucoma Medications: A Randomized Clinical Trial
Brief Title: Visual Function Changes After Intraocular Pressure Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP 1021/05
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Glaucoma
Keywords: intraocular pressure; contrast sensitivity; visual function
MeSH Terms: conditions — Glaucoma

INTERVENTIONS:
Drug: timolol maleate 0,5%
Drug: brimonidine tartrate 0,2%
Drug: travoprost 0,004%

SUMMARY:
During the glaucomatous disease process, subpopulations of cells may be dead, damaged or healthy. Visual function changes could be observed due to a recovering of the suffering ganglion cells after the intraocular pressure reduction. This study aims at evaluating the correlation between intraocular pressure reduction and visual function changes in glaucoma patients after using antiglaucoma medications.

DETAILED DESCRIPTION:
Primary open angle glaucoma patients without use of antiglaucoma medications will be enrolled in this study. After inclusion, the patients will randomly receive one of three antiglaucoma medications (timolol maleate 0,5%, brimonidine tartrate 0,2% or travoprost 0,004%) in one randomly selected eye.

The patients will be evaluated with Goldmann applanation tonometry, visual acuity test, contrast sensitivity test, visual quality perception test (visual analogue scale) and standard automated perimetry before and after 4 weeks of glaucoma treatment onset.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Intraocular pressure greater than 21 mmHg

Exclusion Criteria:

* Best corrected visual acuity (BCVA) worse than 20/80
* Significant media opacity
* History of steroid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
intraocular pressure
contrast sensitivity
visual quality perception

SECONDARY OUTCOMES:
Mean deviation of the visual field (MD)
Pattern Standard Deviation of the visual field (PSD)
visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Prata, MD, Principal Investigator — Federal University of São Paulo; Luiz A Melo Jr, MD, Principal Investigator — Federal University of São Paulo